CLINICAL TRIAL: NCT04652388
Title: The Impact of Nutritional Counselling in Children With Autistic Spectrum Disorder
Brief Title: Impact of Nutritional Counselling in Children With Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, Chief of the Pediatric Allergy Program at the Department of Translational Medical Science Chief of the ImmunoNutritionLab at CEINGE - Advanced Biotechnologies, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 353/20
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional counseling (Experimental): Children with autism spectrum disorders to whom administer nutritional counseling
  Interventions: Behavioral: Nutritional counseling
- Controls (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Nutritional counseling — Nutritional counseling about mediterranean diet
  Arms: Nutritional counseling

SUMMARY:
Autism Spectrum Disorder (ASD) is a complex group of behavioral disorders characterized by defects in social interaction and communication associated with restricted and repetitive behaviors and activities. The prevalence in pediatric age is continuously increasing in Western countries (58-67 / 10,000). The Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) describes a worldwide population prevalence of approximately 1%. According to the latest data from the National Observatory for the monitoring of ASD, in Italy 1 child out of 77 (age 7-9 years) has the disease with a higher prevalence in males: males are affected 4.4 times more than females . The clinical manifestations of ASD are the result of complex interactions between genetic, epigenetic, environmental and microbiological factors. Alterations in nutritional status, eating habits and adverse reactions to food appear to be more frequent in children with ASD. It is estimated that 46-89% of children with ASD have feeding problems which can include unusual eating patterns, rituals and food selectivity. These types of eating behaviors can lead to severe alterations in nutritional status. Furthermore, the data present in the literature concerning the eating habits of children with ASD suggest a high consumption of "junk food" and foods rich in calories together with a refusal of fruit, vegetables or proteins. These data suggest that the dietary and behavioral problems frequently present in these children could favor a condition of obesity. Finally, a high percentage of children with ASD undergo elimination diets, characterized by exclusions of foods relevant to the diet of a child such as milk and gluten to alleviate the symptoms of the disease. Such elimination diets are only rarely supervised by a nutritionist with further consequences on nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autism spectrum disorders

Exclusion Criteria:

* Age at enrollment <24 or> 48 months.
* Concomitant presence of other chronic diseases
* epilepsy,
* neurological syndromes,
* immunodeficiencies,
* diabetes,
* congenital heart disease,
* autoimmune diseases,
* inborn errors of metabolism,
* tuberculosis,
* cystic fibrosis,
* chronic respiratory tract diseases,
* inflammatory bowel disease,
* celiac disease,
* eosinophilic pathologies of the gastrointestinal tract,
* functional gastrointestinal disorders,
* obesity,
* tumors,
* malnutrition • Major malformations or previous surgery of the gastrointestinal / urinary / respiratory tract.

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Mediterranean Diet | change from baseline at 12 months
  Evaluation of mediterranea diet through score aiming to assess the mediterranean diet adhesion (Kidmed score; minimum value 0-worse maximum value 12-better)

SECONDARY OUTCOMES:
Change in food selectivity | change from baseline at 12 months
  Evaluation of Food Preferences Inventory score (cut off 47; <47 selective child)
Change in eating habits | change from baseline at 12 months
  Evaluation of 3-day diary foods

OTHER OUTCOMES:
change in auxological parameters | change from baseline at 12 months
  Evaluation of body growth, height

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided